CLINICAL TRIAL: NCT01802814
Title: International Study for Treatment of Standard Risk Childhood Relapsed ALL 2010 A Randomized Phase III Study Conducted by the Resistant Disease Committee of the International BFM Study Group
Brief Title: International Study for Treatment of Standard Risk Childhood Relapsed ALL 2010
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Australian & New Zealand Children's Haematology/Oncology Group (Other); St. Anna Kinderkrebsforschung (Co-Sponsor Austria) (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network); University Hospital, Motol (Other); Copenhagen University Hospital (Rigshospitalet) (Co-Sponsor Copenhagen) (Unknown); Turku University (Co-Sponsor Finland) (Unknown); Centre Hospitalier Universitaire de Nice (Other); Our Lady's Chilrden's Hospital (Co-Sponsor Ireland) (Unknown); Tel Aviv Sourasky Medical Centre (Co-Sponsor Israel) (Unknown); Ospedale Pediatrico Bambino Gesù (Co-Sponsor Italy) (Unknown); National Hospital Organization Nagoya Medical Center (Co-Sponsor Japan) (Unknown); Prinses Máxima Centrum (Co-Sponsor Netherlands) (Unknown); Oslo University Hospital (Co-Sponsor Oslo) (Unknown); Medical University of Wroclaw (Co-Sponsor Poland) (Unknown); Instituto Português de Oncologia de Lisboa (Co-Sponsor Lisboa) (Unknown); Spanish Society of Pediatric Hematology and Oncology (SEHOP) (Co-Sponsor Spain) (Unknown); University Children's Hospital, Zurich (Other); Central Manchester University (Co-Sponsor United Kingdom) (Unknown)
Responsible Party: Principal Investigator, PD Dr. Arend von Stackelberg, PD Dr. med. Arend von Stackelberg, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IntReALL SR 2010
Record Dates: First submitted 2013-02-18; First posted 2013-03-01 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Receptors, Scavenger; epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SR-A (No Intervention): Patients randomized to the SR-A Arm receive induction, consolidation and maintenance therapy according to a modified protocol ALL-REZ BFM 2002 with Protocol II-IDA as 1st consolidation element. In this arm patients are randomized not to receive epratuzumab.This randomization has been stopped pre-term on 1.2.2019 since the investigational product is not provided anymore by the manufacturer.
- SR-A + Epratuzumab (Active Comparator): Patients randomized to the SR-A Arm receive induction, consolidation and maintenance therapy according to a modified protocol ALL-REZ BFM 2002 with Protocol II-IDA as 1st consolidation element. In this arm patients are randomized to receive epratuzumab. This randomization has been stopped pre-term on 1.2.2019 since the investigational product is not provided anymore by the manufacturer.
  Interventions: Drug: SR-A + Epratuzumab
- SR-B (No Intervention): Patients randomized to the SR-B Arm receive induction, post-induction and maintenance therapy according to the protocol ALL-R3. In this arm patients are randomized not to receive epratuzumab. This randomization has been stopped pre-term on 1.2.2019 since the investigational product is not provided anymore by the manufacturer.
- SR-B + Epratuzumab (Active Comparator): Patients randomized to the SR-B Arm receive induction, post-induction and maintenance therapy according to the protocol ALL-R3. In this arm patients are randomized to receive epratuzumab. This randomization has been stopped pre-term on 1.2.2019 since the investigational product is not provided anymore by the manufacturer.
  Interventions: Drug: SR-B + Epratuzumab

INTERVENTIONS:
Drug: SR-A + Epratuzumab
  Other Names: Epratuzumab
  Arms: SR-A + Epratuzumab
Drug: SR-B + Epratuzumab
  Other Names: Epratuzumab
  Arms: SR-B + Epratuzumab

SUMMARY:
The main goal of this study is to improve the outcome of children and adolescents with standard risk (SR) first relapsed acute lymphoblastic leukemia. Furthermore, goal is to set up a large international study group platform allowing for optimization of standard treatment strategies and integration of new agents.

DETAILED DESCRIPTION:
ALL is the most frequent malignancy in childhood and has favourable event-free and overall survival rates. About 15% of patients suffer relapse. At relapse prognosis is much inferior (about 50% survival) leukemic clones exhibit much more resistance to conventional chemotherapy. Patients with relapse require treatment intensification and different therapeutic strategies. At relapse, new targeted agents can provide the chance for better cure rates and need to be investigated in prospective controlled trials before they may be even eligible for frontline treatment strategies.

The IntReALL SR 2010 trial is designed to achieve 2 major aims: Establishment of the best available standard chemotherapy treatment. This is addressed with the randomization of the 2 best developed strategies for treatment of childhood relapsed ALL, the German ALL-REZ BFM 2002 Protocol with the Protocol II IDA arm, and the British ALL-R3 protocol with the mitoxantrone arm. This randomization allows confirming the feasibility of both protocols in a large variety of different countries and study groups with different frontline therapy strategies. As result from this trial a common standard chemotherapy for childhood relapsed ALL will be developed which can serve as backbone for investigation of the most attractive targeted new agents.

The 2nd aim is the investigation of the efficacy and tolerability of the humanized CD22 directed monoclonal antibody Epratuzumab, manufactured and provided by the company Immunomedics, US. The drug will be randomly added to the respective consolidation chemotherapy, using EFS as primary endpoint. Epratuzumab has been developed in adult rheumatology indications and in B-cell malignancies. A phase I and early phase II combination trial in childhood relapse ALL has been conducted and published by the Children's Oncology Group (COG), and results of an extended phase II trial have been recently presented at the ASH meeting (12/2011). The drug showed a very favourable safety profile as single drug and in combination with multidrug chemotherapy. Activity was moderate, the recent trial showed a significantly better elimination of minimal residual disease (MRD) in patients achieving a 2nd complete remission. This finding supports the strategy to use Epratuzumab in combination with consolidation chemotherapy after induction in patients having reduced the leukemia burden in the bone marrow to at least below 25%, most of them will be in 2nd complete remission. Epratuzumab will be given weekly at the established dose. Pharmacokinetics will be investigated in a reduced number of patients. The further treatment will be conventional intensive chemotherapy and maintenance therapy in patients with good MRD response after induction, or with allogeneic stem-cell transplantation (SCT) in those with insufficient MRD response. SCT will be considered as standard treatment element and will not lead to censoring of the patients of considered as endpoint. Epratuzumab is not licensed so far and the trial may add to the approval process in case.

Scientific advice for the trial has been requested at the FDA and the EMA. Both institutions have responded supportively. Concerns and recommendations of FDA and EMA have been addressed in the protocol and the corresponding statistical analysis plan.

The IntReALL SR 2010 trial will be financed within the FP7 project IntReALL 2010 supported by the European Commission. Within the project next to the SR trial a strategy for high Risk (HR) patients will be addressed, the establishment of harmonized diagnostic procedures, an international tumour bank and a comprehensive biologic/scientific programme will be set up, a web-based Good Clinical Practice (GCP) conform database will be established, a comprehensive statistical strategy for both trials are established, and drug development in this indication will be promoted and organized from side of the disease experts in cooperation with the established academic structures ITCC (Innovative Therapies for Children with Cancer), the ENCCA project (European Network for Cancer in Children and Adolescents) and SIOPe (International Society for Pediatric Oncology Europe), the central authorities (EMA, FDA) and Industry. Parent organisation and former patients are integrated into and accompany the process.

Main aims of the IntReALL FP7 project are to establish a therapeutic platform for children with relapsed ALL in Europe and beyond and to give them access to the most promising new agents under academic control and free from commercial interests.

Randomized evidence for efficacy and tolerability of new drugs are demanded by competent authorities. These trials are conducted beyond the mostly palliative patient group eligible for phase I/II trials in curative indications. Treatment protocols for with curative indications need to be conducted in the best interests of the patients, ideally with an academic sponsor. The design should be driven by medical and scientific evidence and not by commercial interests as is the case in industry sponsored trials. This concept was acknowledged by the European Commission selecting the project for funding from many other powerful applications.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed diagnosis of 1st relapsed precursor B-cell or T-cell ALL
* Children less than 18 years of age at inclusion
* Meeting SR criteria: late isolated or late/early combined B-cell precursor (BCP) bone marrow (BM) relapse, any late/early isolated extramedullary relapse
* Patient enrolled in a participating centre
* Written informed consent
* Start of treatment falling into the study period
* No participation in other clinical trials 30 days prior to study enrolment that interfere with this protocol, except trials for primary ALL Inclusion criteria specific for the epratuzumab randomization
* Precursor B-cell immunophenotype. A specific CD22 expression level is not required
* M1 or M2 status of the bone marrow after induction

Exclusion Criteria:

* BCR-ABL / t(9;22) positive ALL
* Pregnancy or positive pregnancy test (urine sample positive for β-HCG > 10 U/l)
* Sexually active adolescents not willing to use highly effective contraceptive method (pearl index <1) until 2 years after end of antileukemic therapy
* Breast feeding
* Relapse post allogeneic stem-cell transplantation
* The whole protocol or essential parts are declined either by patient himself/herself or the respective legal guardian
* No consent is given for saving and propagation of pseudonymized medical data for study reasons
* Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion (e.g. malformation syndromes, cardiac malformations, metabolic disorders)
* Karnovsky / Lansky score < 50%
* Subjects unwilling or unable to comply with the study procedures
* Subjects who are legally detained in an official institute

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
SR induction/consolidation ALL-REZ BFM 2002 versus UK-ALL-R3 (randomisation 1) | Up to 9 years
  SR induction/consolidation ALL-REZ BFM 2002 versus UK-ALL-R3 (randomisation 1): 10% pEFS superiority of arm B above a 65% pEFS at 4 years of arm A
SR consolidation +/- epratuzumab (randomisation 2) | Up to 9 years
  SR consolidation +/- epratuzumab (randomisation 2): 10% pEFS superiority of the arm with epratuzumab above an expected 74% pEFS at 4 years of the standard arm

SECONDARY OUTCOMES:
SR induction/consolidation | Up to 9 years
  SR induction/consolidation: comparison of OS, toxicity, rate of CR2, and rate of MRD between treatment groups
SR consolidation +/- epratuzumab | Up to 9 years
  SR consolidation +/- epratuzumab: comparison of OS, toxicity, MRD levels, rate of MRD and evaluation of pharmacokinetic parameters of Epratuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Arend von Stackelberg, MD, Principal Investigator — University Hospital of Berlin - Charité
Locations (17):
- Australian & New Zealand Childhood Hematology & Oncology Group, Clayton, Victoria, Australia
- St. Anna Kinderkrebsforschung, CCRI, Vienna, Austria
- Hòpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium
- University Hospital Motol, Prague, Czechia
- Copenhagen University Hospital (Rigshospitalet), Copenhagen, Denmark
- Turku University Central Hospital, Turku, Finland
- CHU Nice, Nice, France
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Tel Aviv Sourasky Medical Centre, Tel Aviv, Israel
- Ospedale Pediatrico Bambino Gesù, Roma, Italy
- St.Lukes International Hospital, Tokyo, Japan
- Prinses Máxima Centrum, Lundlaan, Utrecht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Dpt. SCT and Hematology/Oncology University Wroclaw, Wroclaw, Poland
- Instituto Português de Oncologia de Lisboa, Lisbon, Portugal
- University Children's Hospital Zurich, Zurich, Switzerland
- Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- See also: Public Website of the FP7 Collaborative Project "IntReALL" — http://www.intreall-fp7.eu/